CLINICAL TRIAL: NCT03062436
Title: Stopping Imatinib Therapy in CML Patients With Sustained Molecular Remission
Brief Title: To Study the Impact of Stopping Therapy in Patients of CML With Molecular Remission
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Command Hospital, India (Other Government)
Responsible Party: Principal Investigator, Sanjeevan Sharma, Clinical Hematologist, Command Hospital, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFMRC 4714/2016
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Chronic Myeloid Leukemia; Treatment Free Remission
Keywords: CML, treatment free remission
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sustained molecular remission (Experimental): Patients of CML who remain in sustained molecular remission at 12 months after Stopping the standard drug therapy
  Interventions: Other: Stopping the standard drug therpy; Diagnostic Test: Quantitative bcrabl recording every month for first 6 months

INTERVENTIONS:
Other: Stopping the standard drug therpy — Stopping the standard drug therapy of CML patients and monitoring their treatment free remission status
Diagnostic Test: Quantitative bcrabl recording every month for first 6 months — Monthly recording of quantitative bcrabl by RQPCR on patients peripheral blood derived RNA. RQPCR will have minimum sensitivity of log4.5

SUMMARY:
Patients with chronic myeloid leukemia (CML) are conventionally put on life long therapy with tyrosine kinase inhibitor drugs (Imatinib mesylate in India). Patients who achieve a deep molecular response which has been sustained for at least three years, can be taken off the drug therapy. Thereafter a close monitoring is required to monitor their disease relapse. In case there is evidence of disease recurrence on highly sensitive molecular assays, their drug therapy is restarted. The study aims to identify proportion of patients who can be kept off drug therapy in a state of sustained molecular remission.

DETAILED DESCRIPTION:
While a large number of studies which have stopped TKI therapy in similar patients exist in Europe and USA, no such study has been done on Indian or other south Asian population. Almost all studies done previously have noted that in relapsed patients, who show disease recurrence on stopping their TKI therapy, their remission state is regained once the TKI therapy is restarted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of CML on TKI (Imatinib) therapy for more than 5 years
2. Patients who have been in complete molecular response (MR 4.5 +) for at least three years

Exclusion Criteria:

1. Patients who ever had blast crisis
2. Patients achieving molecular response with second generation TKI due to failure of Imatinib

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease Recurrence | 12 months from cessation of the drug therapy
  Re-appearance of bcr-abl transcripts by RQPCR at a level >0.01%

CONTACTS AND LOCATIONS:
Locations (1):
- Command Hospital, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No